CLINICAL TRIAL: NCT04092777
Title: 1/2 Building Infrastructure for Community Capacity in Accelerating Integrated Care and 2/2 Building Infrastructure for Community Capacity in Accelerating Integrated Care
Brief Title: Building Infrastructure for Community Capacity in Accelerating Integrated Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, Margarita Alegria, PhD, Chief, Disparities Research Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P002918
Record Dates: First submitted 2019-08-14; First posted 2019-09-17 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Mental Health
Keywords: ACOs; Medicaid; Racial; Ethnic; Linguistic; Minorities
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strong Minds Program (Experimental): This is a 10-session, culturally-adapted intervention, that includes cognitive behavioral therapy techniques combined with mindfulness exercises, led by a Community Health Worker.
  Interventions: Behavioral: Strong Minds
- Enhanced Usual Care (Other): Enhanced usual care includes check in calls by a Care Manager 4 times over the course of 6 months and educational materials about depression and anxiety.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Strong Minds — The proposed intervention integrates cognitive behavioral therapy techniques combined with mindfulness exercises and promotion of behavioral activation through pleasant activities and developing supportive relationships. The intervention is led by CHWs and organized into 10 sessions, tailored to the participant using a collaborative approach, to improve mood symptoms, augment self-reported functioning, and increase self-reported quality of care among participants with moderate to severe symptoms of depression and/or anxiety. It is complemented by a care manager that links participant to services for needs related to social determinants of health (i.e. education, housing). The intervention has been tailored for delivery by CHWs in Spanish, Mandarin, Cantonese, and English.
  Arms: Strong Minds Program
Other: Enhanced Usual Care — Participants in this arm will receive a booklet about anxiety and depression in Spanish, English, or Mandarin/Cantonese. The Care Manager will call the participant 4 times over the course of 6 months to administer the PROMIS depression (8 item) and anxiety (7 item) short forms, a suicide questionnaire, and a question about medication side effects to mimic the administration schedule in the intervention group. With patient's permission, the care manager will inform the PCP about screening and other assessments and determine if participants should be referred to mental health or substance services and removed from control group given symptom severity.
  Arms: Enhanced Usual Care

SUMMARY:
Although the Affordable Care Act (ACA) expanded Medicaid eligibility, Medicaid expansions do not appear to have decreased the gap in mental health treatment between Whites and racial/ethnic or linguistic minorities. There is a critical shortage of trained providers who can offer culturally congruent mental health service in non-English languages in Medicaid-based Accountable Care Organizations (ACOs). Building capacity and training opportunities to implement evidence-based mental health interventions by community health workers (CHWs) could expand ACOs infrastructure and increase access to and quality of mental healthcare. To this end, the investigators will test the effectiveness and implementation of the STRONG MINDS model to improve engagement and quality of treatment for depression and anxiety among low-income racial/ethnic and linguistic minority populations, served by Medicaid ACOs. Our proposed study is a Hybrid Type I Effectiveness Implementation study of the effectiveness of the mental health intervention and its impact on study outcomes within varying contexts associated with Medicaid ACOs in North Carolina (NC) and Massachusetts (MA).

DETAILED DESCRIPTION:
The investigators will test the STRONG MINDS intervention with adults who have moderate to severe symptoms of depression or anxiety, originally defined as 66+ on the CAT-MH for depression and/or 51+ on the CAT-MH for anxiety. Based on psychometric analyses conducted by the developer of the CAT, Dr. Robert Gibbons has two times adjusted the depression and anxiety thresholds to best map onto moderate symptoms for diverse language groups. As of 10/4/19, the criteria for depression had been changed to a cut-off of 50+ on the CAT-MH depression screener or a positive on the CAT-MH for Major Depressive Disorder (MDD is a positive/negative measure, not a dimensional severity score). As of 12/2020, psychometric analysis showed differences across language groups in symptom severity, and the cut offs were updated to include participants who scored 50+ on the CAT-MH depression in English; a score of 42+ for the CAT-MH depression administered in Spanish or in Chinese. Similarly, the developer of the CAT-MH also changed the cut-off scores for anxiety, with 51+ for the CAT-MH anxiety administered in English; but a score of 41+ for the CAT-MH administered in Spanish or Chinese. The MDD remains a positive/negative item at the same thresholds. These analysis and updates help ensure that the adaptive screener is optimally calibrated to diverse language samples. Eligible participants cannot be receiving mental health care (therapy sessions with psychiatrist, psychologist or social worker) in the past 3 months or in the upcoming month. Participants must speak English, Spanish, Mandarin, or Cantonese. Eligible participants will be consented and assigned to a CHW within the site. After a baseline interview, participants will be randomized to either the intervention or an enhanced usual care condition. Randomization will be stratified by site using a computer-generated block randomization scheme of variable block size. The investigators will monitor engagement in treatment (% of participants with 2 or more mental health sessions/visits in a 6-month period after baseline), mental health symptoms (HSCL-25), overall functioning (WHODAS 2.0), and participant perceived quality of care (PoC) for the intervention group and compare to the enhanced control group. Outcome measures (identified above) will be assessed four times during the study period: at baseline, 3 months, 6 months and 12 months.

Recruitment Strategy: CHWs will screen 6,000 participants with the CAT-MH and substance use measures (for exclusion) in addition to obtaining demographic and social determinants information during the 3.5 years of study screening to identify approximately 1,200 eligible participants across both MA and NC (600 per site). Eligible participants will be randomized to the intervention or enhanced control condition and be invited to complete a baseline assessment as described above. Based on data from our clinical trials, the investigators anticipate that 30-33.5% of those screened will show moderate to severe symptoms of depression and/or anxiety and will not be receiving mental health care. The investigators conservatively anticipate that 60-70% will agree to participate, for approximately 600 cases per site with 20% attrition over a 6 month period.

Sampling, Recruitment and Consent: Community Health Workers (CHWs) and Research Assistants (RAs) will be responsible for approaching potential participants in designated clinics or Community-based Organizations (CBOs). In clinics, CHWs will recruit in waiting rooms or by provider referrals. In community agencies, they will recruit during special community events and meetings. Eligible patients will be scheduled for a baseline interview with a Research Assistant that includes instruments designed to identify elevated mental health symptoms, as well as socio-demographics, cultural, contextual and social factors, medication use, health literacy, language proficiency, past access to health services, migration, patient activation and self-management, and motivation to enter care. Following the baseline interview, participants will be randomized to either the intervention or enhanced usual care (control) condition. Additional interviews will be administered by research assistants blind to study condition at 3-, 6- and 12-months following baseline.

ELIGIBILITY:
Inclusion Criteria:

* Latino, Asian, Black (African American or Afro-Caribbean), or non-Latino White
* Adult 18+
* Moderate to severe depressive or anxiety symptoms
* Speak English, Spanish, Mandarin, or Cantonese.

Exclusion Criteria:

* history of psychosis, mania, or psychotic symptoms according to items from the IMPACT study
* self-reported receipt of specialty mental health treatment within past 3 months or upcoming behavioral health appointment in the next month (pharmacological treatments are not excluded)
* evidence that the patient lacks capacity to consent (measured by a validated screener)
* evidence of current suicidal risk or harm to others (affirmative responses on Paykel suicide questionnaire);
* severe alcohol or substance dependence as defined by score of 70+ on the CAT-SA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Alegria, Ph.D., Principal Investigator — Massachusetts General Hospital; Gabriela Livas Stein, Ph.D., Principal Investigator — University of North Carolina, Greensboro
Locations (2):
- United States (2):
  - South Cove Community Health Center, Quincy, Massachusetts
  - MGH Broadway Primary Care - Revere, Revere, Massachusetts

REFERENCES:
- [Derived] Alegria M, Stein GL, Cruz-Gonzalez M, Falgas-Bague I, Markle SL, Eddington KM, Supple A, Fuentes L, Poindexter C, Shrout PE. Building community capacity in mental health care with the Strong Minds-Strong Communities programme: a randomised controlled trial in the USA. Lancet. 2025 Aug 23;406(10505):832-845. doi: 10.1016/S0140-6736(25)00859-1. PMID 40849140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Staff recruited participants from 20 community based organizations and 17 clinics serving a high proportion of clients who identify as Latino (primarily Spanish speaking), Asian (mainly Mandarin or Cantonese speaking), or Black (primarily English speaking). Half of the participants were recruited in North Carolina and half in Massachusetts. From September 4, 2019, to March 2, 2023, research staff assessed 2,584 potential participants for eligibility.
Pre-assignment Details: No significant events in the study occurred after participant enrollment.
Period: Overall Study
Arm/Group | Strong Minds Program | Enhanced Usual Care
Started | 524 | 520
Completed | 488 | 469
Not Completed | 36 | 51
Not completed — Lost to Follow-up | 28 | 46
Not completed — Withdrawal by Subject | 8 | 5

BASELINE CHARACTERISTICS:
Population: Analysis population followed intent-to-treat principles and included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Strong Minds Program | Enhanced Usual Care | Total
Number analyzed (Participants) | 524 | 520 | 1044
Age, Continuous [Mean (Standard Deviation); unit: years] — Self-reported age in years
  years | 42.4 (13.2) | 42.8 (13.4) | 42.6 (13.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 77 | 88 | 165
  Gender: Female | 446 | 429 | 875
  Gender: Other | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and ethnicity: Non-Latino White | 46 | 46 | 92
  Race and ethnicity: Non-Latino Black | 69 | 80 | 149
  Race and ethnicity: American Indian | 2 | 1 | 3
  Race and ethnicity: Non-Latino Asian | 69 | 68 | 137
  Race and ethnicity: Latino | 332 | 322 | 654
  Race and ethnicity: Mixed | 4 | 3 | 7
  Race and ethnicity: Other | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Massachusetts | 263 | 259 | 522
  United States: North Carolina | 261 | 261 | 522
Hopkins Symptom Checklist-25 (HSCL-25) [Mean (Standard Deviation); unit: units on a scale] — The Hopkins Symptom Checklist-25 (HSCL-25) is a 25-item measure of self-reported depression and anxiety symptoms in the past two weeks rated on a 4-point scale from 1 'not at all' to 4 'extremely'. Total scores are calculated as the average of all items (range 1 to 4), where higher scores represent worse depression and anxiety symptoms.
  units on a scale | 2.1 (.5) | 2.1 (.5) | 2.1 (.5)
World Health Organization Disability Assessment Schedule 2.0 [Mean (Standard Deviation); unit: units on a scale] — The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) is a 12-item self-reported measure of level of functioning in six domains: cognition, mobility, self-care, getting along, life activities, and participation. Participants rate difficulties performing activities in each domain in the past 30 days using a 5-point scale from 1 'none' to 5 'extremely or cannot do'. Total scores are calculated as the sum of all items (12 to 60), with higher scores indicating lower functioning levels.
  units on a scale | 23.8 (8.9) | 23.3 (8.6) | 23.5 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Engagement in Mental Health Intervention Sessions
Description: Engagement in Mental Health Intervention Sessions was measured as attending 2 or more (out of 10) sessions of STRONG MINDS. This outcome was measured among intervention participants only (Strong Minds Program) using an indicator variable equal to one if a participant attended 2+ intervention sessions, and equal to zero otherwise.
Time Frame: 6 months after baseline
Population: Analysis followed intent-to-treat principles and included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Strong Minds Program | Enhanced Usual Care
Number analyzed (Participants) | 524 | 0
Participants | 464 |

2. Primary Outcome: Hopkins Symptoms Checklist-25; HSCL-25 (Change)
Description: The Hopkins Symptom Checklist-25 (HSCL-25) is a 25-item measure of self-reported depression and anxiety symptoms in the past two weeks rated on a 4-point scale from 1 'not at all' to 4 'extremely'. Total scores are calculated as the average of all items (range 1 to 4), where higher scores represent worse depression and anxiety symptoms.
Time Frame: Baseline, 3 months, 6 months, and 12 months after baseline
Population: Analysis followed intent-to-treat principles and included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Strong Minds Program | Enhanced Usual Care
Number analyzed (Participants) | 524 | 520
score on a scale
  Scores at month 3 adjusted for baseline scores | 1.65 (0.02) | 1.84 (0.02)
  Scores at month 6 adjusted for baseline scores | 1.61 (0.02) | 1.81 (0.02)
  Scores at month 12 adjusted for baseline scores | 1.64 (0.02) | 1.78 (0.02)

3. Primary Outcome: Functioning: WHODAS 2.0 (Change)
Description: The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) is a 12-item self-reported measure of level of functioning in six domains: cognition, mobility, self-care, getting along, life activities, and participation. Participants rate difficulties performing activities in each domain in the past 30 days using a 5-point scale from 1 'none' to 5 'extremely or cannot do'. Total scores are calculated as the sum of all items (12 to 60), with higher scores indicating lower functioning levels.
Time Frame: Baseline, 3 months, 6 months, and 12 months after baseline
Population: Analysis followed intent-to-treat principles and included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Strong Minds Program | Enhanced Usual Care
Number analyzed (Participants) | 524 | 520
score on a scale
  Scores at 3 months adjusted for baseline scores | 19.91 (0.34) | 21.42 (0.32)
  Scores at 6 months adjusted for baseline scores | 19.01 (0.36) | 21.50 (0.35)
  Scores at 12 months adjusted for baseline scores | 19.74 (0.39) | 21.46 (0.35)

4. Primary Outcome: Perceptions of Care Outpatient Survey (PoC-OP) (Change)
Description: Perceived quality of care was measured using the Global Evaluation of Care domain of the Perceptions of Care Outpatient Survey (PoC-OP), a clinical-care oriented, self-report satisfaction rating scale assessing patients' perception of the quality of interpersonal care. The Global Evaluation of Care domain includes three items rated on a 4-point scale from 1 'never' to 4 'always', transformed into a score from 0 'lowest quality' to 100 'highest quality'.
Time Frame: Baseline, 3 months, 6 months, and 12 months after baseline
Population: Analysis followed intent-to-treat principles and included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Strong Minds Program | Enhanced Usual Care
Number analyzed (Participants) | 524 | 520
score on a scale
  Scores at 3 months | 87.00 (1.02) | 74.44 (1.02)
  Scores at 6 months | 86.37 (1.11) | 77.72 (0.93)
  Scores at 12 months | 83.15 (0.98) | 76.71 (1.00)

5. Secondary Outcome: CAT-MH Depression (Change)
Description: Computerized Adaptive Test for Mental Health (CAT-MH), is a suite of validated computer adaptive tests. CAT-MH scores are based on responses to algorithm-selected items that minimize participant burden using item response theory methodology. The adaptive nature of the CAT-MH targets a participant's specific level of severity at that point in time. The number of items at each time point varies because the same questions are not repeatedly administered. The depression subscale assesses severity of depressive symptoms. Total scores range from 0 to 100 with higher scores indicating worse depression symptoms.
Time Frame: Baseline, 3 months, 6 months, and 12 months after baseline
Population: Analysis followed intent-to-treat principles and included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Strong Minds Program | Enhanced Usual Care
Number analyzed (Participants) | 524 | 520
score on a scale
  Scores at month 3 adjusted for baseline scores | 39.06 (0.80) | 46.34 (0.78)
  Scores at month 6 adjusted for baseline scores | 37.99 (0.90) | 45.66 (0.85)
  Scores at month 12 adjusted for baseline scores | 39.74 (0.92) | 45.19 (0.83)

6. Secondary Outcome: CAT-MH Anxiety (Change)
Description: Computerized Adaptive Test for Mental Health (CAT-MH), is a suite of validated computer adaptive tests. CAT-MH scores are based on responses to algorithm-selected items that minimize participant burden using item response theory methodology. The adaptive nature of the CAT-MH targets a participant's specific level of severity at that point in time. The number of items at each time point varies because the same questions are not repeatedly administered. The anxiety subscale assesses severity of anxiety symptoms. Total scores range from 0 to 100 with higher scores indicating worse anxiety symptoms.
Time Frame: Baseline, 3 months, 6 months, and 12 months after baseline
Population: Analysis followed intent-to-treat principles and included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Strong Minds Program | Enhanced Usual Care
Number analyzed (Participants) | 524 | 520
score on a scale
  Scores at month 3 adjusted for baseline scores | 32.82 (0.93) | 40.06 (0.85)
  Scores at month 6 adjusted for baseline scores | 31.08 (1.00) | 39.61 (1.01)
  Scores at month 12 adjusted for baseline scores | 33.48 (0.96) | 37.70 (0.97)

ADVERSE EVENTS:
Time Frame: 12 months
Description: We considered as an adverse event the report of a 5 (a suicide attempt) on the Paykel suicidality screener after enrollment. We also considered cases where a participant passed away during the trial.
Arm/Group | Strong Minds Program | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/524 | 2/520
Serious Adverse Events (participants affected / at risk) | 3/524 | 4/520
Other Adverse Events (participants affected / at risk) | 0/524 | 0/520
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Strong Minds Program (N=524) | Enhanced Usual Care (N=520)
Report of a 5 (a suicide attempt) on the Paykel suicidality screener after enrollment (Psychiatric disorders) | 3 | 4

LIMITATIONS AND CAVEATS:
The study was concluded as planned and no technical problems with measurement were experienced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT04092777/Prot_SAP_000.pdf